CLINICAL TRIAL: NCT02132819
Title: The Effect of Withholding Feeds During Red Blood Cell Transfusion on Development of TRAGI in Very Low Birth Weight Infants
Brief Title: Withholding Feeds During Red Blood Cell Transfusion and TRAGI
Acronym: Tx-TRAGI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zekai Tahir Burak Women's Health Research and Education Hospital (Other)
Responsible Party: Principal Investigator, Suzan Sahin, Fellow in Neonatology, Pediatrician, Zekai Tahir Burak Women's Health Research and Education Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Sahin1
Record Dates: First submitted 2014-04-17; First posted 2014-05-07 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2014-05

CONDITIONS: Transfusion; Feeding During Transfusion; Transfusion Related Acute Gut Injury; Necrotising Enterocolitis
Keywords: transfusion; feeding; TRAGI; NEC
MeSH Terms: conditions — Enterocolitis, Necrotizing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Feeding During Transfusion (Placebo Comparator): The feeding process will be continued during the transfusion
  Interventions: Other: feeding during transfusion
- witholding feeds (Active Comparator): At least 2 feeds before the transfusion, 2 feeds after the transfusion and feeds during the transfusion are withholded
  Interventions: Other: Withholding feeds

INTERVENTIONS:
Other: Withholding feeds — At least 2 feeds before the transfusion, 2 feeds after the transfusion and feeds during the transfusion are withholded
  Arms: witholding feeds
Other: feeding during transfusion — The feeding process will be continued during the transfusion
  Arms: Feeding During Transfusion

SUMMARY:
Necrotising enterocolitis (NEC) is a devastating picture that all the neonatologists are afraid of facing during the follow up of newborns. During the last years, investigators ran retrospective observational studies abut NEC developing within the 48 hours after red blood cell transfusion. In the previous studies, the incidence of transfusion associated NEC (TANEC) was found to be 20-35%.Multiple transfusions potentially cause an increased risk for retinopathy of prematurity (ROP) and NEC. Investigators have also proposed a hypothesis about transfusion related acute gut injury (TRAGI), an adverse reaction of transfusion, similar to transfusion related acute lung injury (TRALI) seen in adults.In most of the neonatology clinics, withholding feeds during transfusion is not preferred. But several recent studies show an increase in the incidence of TANEC if the newborn goes on feeding before, during and after the transfusion process, especially if it is fed with a formula. The main aim of this study is to investigate the effect of withholding feeds during transfusion, on the development of TRAGI.

ELIGIBILITY:
Inclusion Criteria:

* <32 weeks of gestational age or <1500 gr, >7 days old premature babies.
* Babies which are fed enterally well at the time of tha planning of transfusion.

Exclusion Criteria:

* Babies with severe sepsis signs.
* Babies with severe hypoxia and asphyxia.
* Babies with congenital anomaly or complex cardiac anomaly.

Ages: 7 Days to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2014-02; Primary Completion 2015-01 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
increase in the abdominal circumference | within 3 days after transfusion but participants will be followed for the duration of hospital stay, an expected average of 5 weeks
  Bell's stage 1/Suspected disease:
  Mild systemic disease (apnoea, bradycardia, temperature instability) Mild intestinal signs (abdominal distention, gastric residuals, bloody stools) Non-specific or normal radiological signs
  Bell's stage 2/Definite disease:
  Mild to moderate systemic signs Additional intestinal signs (absent bowel sounds, abdominal tenderness) Specific radiologic signs (pneumatosis intestinalis or portal venous air) Laboratory changes (metabolic acidosis, thrombocytopaenia)
  Bell's stage 3/Advanced disease:
  Severe systemic illness (hypotension) Additional intestinal signs (striking abdominal distention, peritonitis) Severe radiologic signs (pneumoperitoneum) Additional laboratory changes (metabolic and respiratory acidosis, disseminated intravascular coagulation)

SECONDARY OUTCOMES:
increase in the amounts of gastric residual aspirates | Within 3 days after the transfusion

OTHER OUTCOMES:
occult or obvious blood in stool | within 1 day after transfusion

CONTACTS AND LOCATIONS:
Overall Officials: Suzan Sahin, MD, Principal Investigator — Zekai Tahir Burak Women's Health Research and Education Hospital
Locations (1):
- Suzan Sahin, Ankara, Altındag, Turkey (Türkiye)